CLINICAL TRIAL: NCT04030858
Title: The INFINITE Study: A Prospective Investigation of a Nutrient-dense Diet in Early Addiction Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northern Arizona University (Other)
Responsible Party: Principal Investigator, Jay Sutliffe, Associate Professor, Northern Arizona University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1410688
Record Dates: First submitted 2019-06-05; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Mental Health Issue; Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Diet, Plant-Based; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with an intervention and control group comparison.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group will eat a nutrient-dense plant-based diet and attend weekly nutrition education sessions.
  Interventions: Behavioral: Plant-based diet + nutrition education
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Plant-based diet + nutrition education — The intervention group will adopt a nutrient-dense dietary pattern and receive nutrition education sessions specific to that lifestyle. The diet protocol is comprised of minimally-processed plant foods such as fruits, vegetables, legumes, beans, nuts and seeds. No refined sugars, added salt, or oil will be included. Dietary fat intake limited to 20% of total calories or less per day. Animal products will be eliminated. This dietary pattern is expected to improve resilience, mood, inflammation, microbiome, spirituality, and overall general health (as measured by weight, cholesterol, blood pressure). The treatment group will also receive weekly nutrition education sessions to support the diet.
  Arms: Treatment group

SUMMARY:
The trial will be placed within an ongoing addiction recovery program at Infinite Recovery in Austin, TX. Members with any addiction enrolling in an inpatient treatment program at Infinite Recovery will be recruited into this 1-year study to evaluate the effectiveness of a plant-based diet to aid drug and/or alcohol addiction recovery. Volunteers willing to participate in the trial will be randomly assigned to a treatment or control group. Those in the treatment group will follow the standard protocol offered by Infinite Recovery, with the exception that they will be provided with only plant-based meals. Both groups will also receive nutrition education to support their dietary plan. Several health and wellbeing endpoints will be assessed as part of the standard care at Infinite Recovery, combined with a few additional measurements described within this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Entering inpatient treatment at Infinite Recovery Addiction Treatment Facility

Exclusion Criteria:

* Pregnant
* Psychiatrically unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-09-03 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Resilience | Change from baseline to week 3
  Measured by the Connor-Davidson Resilience Scale (CD-RISC); scale scores range 0-100, with higher values representing better outcomes.
Resilience | Change from baseline to week 10
  Measured by the Connor-Davidson Resilience Scale (CD-RISC); scale scores range 0-100, with higher values representing better outcomes.

IPD SHARING:
Plan to Share IPD: No